CLINICAL TRIAL: NCT06210932
Title: Effects of Social, Emotional and Ethical Development Curriculum (SEED) Video Intervention on Preschoolers: A Randomized Controlled Trial
Brief Title: Social Emotional and Ethical Development (SEED) Video Curriculum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Winnie W.S. MAK, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SBRE-23-0422
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Development, Child; Mindfulness
Keywords: social and emotional skills development; early childhood
MeSH Terms: interventions — Seeds

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group-seed video (Experimental): The participants will engage in a total of four weeks of intervention. The intervention sessions are conducted three times per week, there will be a total of 12 intervention sessions. The intervention group will receive a social, emotional, and ethical development video intervention. They will watch three videos per week for a total of four weeks. The videos will be designed to promote social, emotional, and ethical development.
  Interventions: Behavioral: Social, Emotional, and Ethical Development (SEED) curriculum videos
- Control group-languag enhancement video (No Intervention): The participants will engage in a total of four weeks of intervention. The intervention sessions are conducted three times per week, there will be a total of 12 intervention sessions. The participants in control group will watch a language enhancement video.

INTERVENTIONS:
Behavioral: Social, Emotional, and Ethical Development (SEED) curriculum videos — In response to fulfilling children's urgent psychosocial needs, the Bodhi Love Foundation (BLF) adapted the Kindness Curriculum for young children in Hong Kong by translating it from English to Chinese and adapting its length and content for implementation in the local kindergarten context. The adapted Kindness Curriculum, renamed as Social, Emotional, and Ethical Development curriculum (SEED), A series of videos are developed based on the SEED curriculum, with specific themes for children in K2 and K3, each video last for approximately 10-12 minutes. They will watch three videos per week for a total of four weeks. The videos will be designed to promote social, emotional, and ethical development.
  Arms: Intervention group-seed video

SUMMARY:
The objectives of the present study are to(1)By implementing the SEED Program and using videos as an intervention, the research aims to enhance these critical skills in young children.(2)The study will be the first of its kind to utilize SEED videos as an intervention for pre-schoolers in Hong Kong.(3)If the intervention proves to be effective, the SEED video project can potentially serve as a pilot program for kindergartens in Hong Kong, introducing more children to the SEED Program and its benefits.

DETAILED DESCRIPTION:
In today's Hong Kong climate of increased focus on children's academic achievement through spoon-fed education, this learning only emphasises children's literacy and subject knowledge. However, "spoon-fed" education is always divorced from the social context, it leads our new generation to be considered as not knowing how to get along with others, lacking emotional management skills, and lacking perseverance and resilience.

Children's social, emotional and moral development are as important as subject knowledge. It is found that children's social-emotional skills can predict their academic performance, more specifically children with higher levels of social-emotional competence show better academic performance, including higher literacy and math scores.

In Hong Kong, most kindergarten curricula are compiled based on the Education Bureau's Kindergarten Education Curriculum Guidelines. Few curricula focus on social, emotional and moral development. Therefore, Bodhi Love Foundation has launched the SEED (Social, Emotional, Ethical Development) Program recently. The SEED Program aims to foster the critical skills for the development of self-awareness, empathy and interconnectedness in young children.

In the post-COVID-19 era of the 21st century, online learning is convenient and students are accustomed to taking video classes at home. Hence, this study will develop a series of videos based on the SEED Program which will serve several purposes: (a) It will become the first study of using SEED video as an intervention for pre-schoolers in Hong Kong (b) It will contribute to our understanding of SEED Video as an intervention, its effect for pre-schooler (c) If the intervention is effective, the SEED video project can become a pilot project for Hong Kong kindergartens to expose more children to SEED.

This study will focus on students in a kindergarten in the North District of Hong Kong, and the results are planned to be expanded to include K2 and K3.

III. Identification of the research problem

1. Does the SEED (Social, Emotional, Ethical Development) video project increase children's social skills?
2. Does the SEED video project enhance the emotional management skills of children?
3. Does the SEED video project improve the executive function of children? IV. Literature Review The most widely used psychological experiments for assessing children's inhibitory has been using structured tests.

The marshmallow test is the most well-known method for assessing children's ability to self-control. In this test, a child is offered a choice between a small immediate reward, such as a marshmallow, or a larger delayed reward, such as two marshmallows, if they can wait for a certain period without eating the initial reward, they can receive the larger delayed reward.

Another widely used task of measuring executive function is the day-night task. In this task, children are required to say the opposite of what they see on the stimulus cards, for instance, say "night" when a white card with the sun is shown and say "day" when a black card with a moon is shown.

The experiments mentioned above were used in this study to achieve a more comprehensive assessment of executive functions in young children. In the marshmallow experiment, stickers will be used as rewards, and an additional component of sharing with others will be included to test children's social skills and willingness to share with others.

In addition, researchers conducted a study to investigate the effectiveness of a video-based social skills training program for developing pre-schoolers. They found that the use of videos is engaging and helpful in promoting social skill development.

V. Research Procedures

The participants in this research study will be K2-K3 pre-schoolers from a kindergarten in Hong Kong. The activities they will engage in include:

Pre-test: Before the intervention begins, the participants will undergo a pre-test to assess their baseline executive function.

Intervention: The participants will be divided into two groups: the intervention group and the control group. The participants will engage in a total of four weeks of intervention. The intervention sessions are conducted three times per week, there will be a total of 12 intervention sessions. The intervention group will receive a social, emotional, and ethical development video intervention. They will watch three videos per week for a total of four weeks. The videos will be designed to promote social, emotional, and ethical development. whereas the control group will receive a language enhancement video intervention.

Post-Test: After the intervention period, both the intervention group and the control group will undergo a post-test to evaluate any changes in their executive function.

Number of Sessions: The participants will engage in a total of four weeks of intervention. The intervention sessions are conducted three times per week, there will be a total of 12 intervention sessions.

Time Commitment: The total time commitment for each participant will depend on the duration of the intervention sessions. Each intervention session lasts approximately 10-12 minutes, the participants will need to allocate approximately 2-2.5 hours over the four-week period.

ELIGIBILITY:
Inclusion Criteria:

- For children: aged 3-7 years old, understand Cantonese

- For parents: aged 18 years old or above, understand Cantonese

Exclusion Criteria:

Unable to understand Cantonese

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 160 (Actual)
Dates: Start 2023-01-20 (Actual); Primary Completion 2024-04-18 (Actual); Study Completion 2024-04-18 (Actual)

PRIMARY OUTCOMES:
Social Skills Improvement System-Rating Scales (Preschool Parents version) (SSIS - SEL) | 4th week
  The Social Skills Improvement System-Rating Scales (Preschool Parents version) consists of 20 items which assess children's skills in each of the five social-emotional learning competencies: Self-Awareness, Self-Management, Social Awareness, Relationship Skills, Responsible Decision Making. Parents indicate answer to the question on 4-point scale ranging from 1 (not at all) to 4(often).
Strengths and Difficulties Questionnaire (SDQ) | 4th week
  A 20-item internalizing and externalizing problems subscales of the Strengths and Difficulties Questionnaire will be used to access their child's adjustment difficulties on a 3-point scale ranging from 1 (not true) to 3 (certainly true). The internalizing problems subscale capture emotional symptoms and peer relationship problems, whereas the externalizing problems subscale capture conduct problems and hyperactivity/inattention.
Delay of Shared Gratification Task | 4th week
  The 5-minute Delay of Shared Gratification Task measures children's sharing behavior involving the small stickers. Children will be asked to share 1-2 stickers with other people over four instances, such as sharing with cost, sharing without cost, and delay of sharing.
Head-Toe-Knees-Shoulders task (HTKS) | 4th week
  The 10-minute Head-Toe-Knees-Shoulders task (HTKS) measures children's behavioral regulation. Specifically, the task requires children to do the opposite of commands. For each command, the experimenter uses a 3-point scale to record the child's responses at 0 = incorrect, 1 = self-correct, and 2 = correct.
Disappointing Gift Task | 4th week
  Disappointing Gift Task measures children's emotion regulation. Specifically, they are informed that they will receive a very nice gift but end up receiving an undesirable gift, e.g., trash paper. Children's facial expression will be observed and coded based on Saarni's emotion coding system.
Children's Behavioral Questionnaire(CBQ) age 3-7 | 4th week
  In the CBQ, parents are asked to rate their child on a 7-point scale ranging from 1 (extremely untrue of your child) to 7 (extremely true of your child). Parents are also provided with a Not Applicable response option when the child has not been observed in the situation described. The standard form consists 15 subscales, in this study, 3 subscales(35 items in total) from standard form are used, namely Attentional Control, Impulsivity and Inhibitory Control.

CONTACTS AND LOCATIONS:
Overall Officials: Winnie WS Mak, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Dept of Psychology, CUHK, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gunter, L., Caldarella, P., Korth, B. B., & Young, K. R. (2012). Promoting social and emotional learning in preschool students: A study of strong start pre-K. Early Childhood Education Journal, 40(3), 151-159. doi:10.1007/s10643-012-0507-z
- [Background] Ling DS, Wong CD, Diamond A. Do children need reminders on the Day-Night task, or simply some way to prevent them from responding too quickly? Cogn Dev. 2016 Jan-Mar;37:67-72. doi: 10.1016/j.cogdev.2015.10.003. PMID 26949287
- [Background] Mischel, W. (2014). The marshmallow test : Mastering self-control. New York: Little, Brown and Company.
- [Background] Shukla-Mehta, S., Miller, T., & Callahan, K. J. (2010). Evaluating the effectiveness of video instruction on social and communication skills training for children with autism spectrum disorders: A review of the literature. Focus on Autism and Other Developmental Disabilities, 25(1), 23-36. doi:10.1177/1088357609352901
- [Background] Blewitt C, Fuller-Tyszkiewicz M, Nolan A, Bergmeier H, Vicary D, Huang T, McCabe P, McKay T, Skouteris H. Social and Emotional Learning Associated With Universal Curriculum-Based Interventions in Early Childhood Education and Care Centers: A Systematic Review and Meta-analysis. JAMA Netw Open. 2018 Dec 7;1(8):e185727. doi: 10.1001/jamanetworkopen.2018.5727. PMID 30646283
- [Background] Bornstein MH, Hahn CS, Haynes OM. Social competence, externalizing, and internalizing behavioral adjustment from early childhood through early adolescence: developmental cascades. Dev Psychopathol. 2010 Nov;22(4):717-35. doi: 10.1017/S0954579410000416. PMID 20883577
- [Background] Collaborative for Academic, Social, and Emotional Learning (CASEL). (2021). CASEL's SEL Framework. https://casel.org/casel-sel-framework-11-2020/
- [Background] Curriculum Development Council, Education Bureau, Hong Kong SAR. (2017). Kindergarten education curriculum guide: Joyful learning through play balanced development all the way.
- [Background] Dunning D, Tudor K, Radley L, Dalrymple N, Funk J, Vainre M, Ford T, Montero-Marin J, Kuyken W, Dalgleish T. Do mindfulness-based programmes improve the cognitive skills, behaviour and mental health of children and adolescents? An updated meta-analysis of randomised controlled trials. Evid Based Ment Health. 2022 Jul 12;25(3):135-42. doi: 10.1136/ebmental-2022-300464. Online ahead of print. PMID 35820989
- [Background] Flook L, Goldberg SB, Pinger L, Bonus K, Davidson RJ. Mindfulness for teachers: A pilot study to assess effects on stress, burnout and teaching efficacy. Mind Brain Educ. 2013 Sep;7(3):10.1111/mbe.12026. doi: 10.1111/mbe.12026. PMID 24324528
- [Background] Flook L, Goldberg SB, Pinger L, Davidson RJ. Promoting prosocial behavior and self-regulatory skills in preschool children through a mindfulness-based Kindness Curriculum. Dev Psychol. 2015 Jan;51(1):44-51. doi: 10.1037/a0038256. Epub 2014 Nov 10. PMID 25383689
- [Background] Heckman, J. J. (2011). The economics of inequality: The value of early childhood education. American Educator, 35(1), 31.
- [Background] Unicef. (2021, October 15). State of the world's children, caring for children's mental health. Retrieved February 15, 2023.
- [Background] World Health Organization. (2018). United Nations Children's Fund, World Bank Group. Nurturing care for early childhood development: a framework for helping children survive and thrive to transform health and human potential. Geneva: World Health Organization. https://apps.who.int/iris/bitstream/handle/10665/272603/9789241514064-eng.pdf